CLINICAL TRIAL: NCT00567840
Title: A Phase IIa Trial to Evaluate the Safety, Tolerability, Extended Early Bactericidal Activity and Pharmacokinetics of 14 Days' Treatment With Four Oral Doses of PA-824 in Adult Participants With Newly Diagnosed, Uncomplicated, Smear-Positive, Pulmonary Tuberculosis
Brief Title: PA-824-CL-007: Phase IIa Evaluation of Early Bactericidal Activity in Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Prof. Andreas Diacon, Tiervlei Trial Center, University of Stellenbosch, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA-824-CL-007
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Early Bactericidal Activity; EBA; pulmonary tuberculosis; PA-824; Pretomanid; CL-007
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — pretomanid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): PA-824 200 mg/qd
  Interventions: Drug: PA-824
- 2 (Experimental): PA-824 600 mg/qd
  Interventions: Drug: PA-824
- 3 (Experimental): PA-824 1000 mg/qd
  Interventions: Drug: PA-824
- 4 (Experimental): PA-824 1200 mg/qd
  Interventions: Drug: PA-824
- 5 (Active Comparator): Rifafour e-275 mg
  Interventions: Drug: PA-824

INTERVENTIONS:
Drug: PA-824 — 200 mg, 600 mg, 100 mg, 1200 mg qd
  Other Names: Rifafour e-275

SUMMARY:
The trial will evaluate the extended bactericidal activity of 14 consecutive days of oral administration of PA-824 at 200, 600, 1000 and 1200 mg per day in adult patients with newly diagnosed, uncomplicated, smear positive tuberculosis. A control group will receive standard TB treatment.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* M/F 18-64 yo
* newly diagnosed pulmonary TB
* sputum positive
* adequate contraception

Exclusion Criteria:

* poor health
* rifampicin resistance
* treatment with other anti TB agents in last 3 mos.
* extrapulmonary TB
* COPD
* neuropathy
* ECG wih QRS prolongation ove 120 msec
* CV disorder
* diabetes requiring insulin
* Metabolic disease
* drug/alcohol abuse
* pregnancy
* use of substances that are strong inhibitors/inducers of CYP450
* use of ARV

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Dawson, MD, Principal Investigator — UCT Lung Institute; Andreas Diacon, MD, Principal Investigator — Tiervlei Trial Center, Stelennbosch University, South Africa
Locations (2):
- South Africa (2):
  - Tiervlei Trials Center, Stellenbosch University, Cape Town, Cape Province
  - University of Cape Town Lung Institute, Cape Town, Cape Province

REFERENCES:
- See also: Related Info — http://www.tballiance.org

RESULTS

PARTICIPANT FLOW:
Groups:
- PA-824 200 mg: PA-824: 200 mg per day for 14 consecutive days
- PA-824 600 mg: PA-824: 600 mg per day for 14 consecutive days
- PA-824 1000 mg: PA-824: 1000 mg per day for 14 consecutive days
- PA-824 1200 mg: PA-824: 1200 mg per day for 14 consecutive days
- Rifafour: Rifafour e-275 on Days 1 to 14, dosed by weight
Period: Overall Study
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Started | 15 | 15 | 16 | 15 | 8
Completed | 13 | 15 | 15 | 14 | 8
Not Completed | 2 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour | Total
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 8 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.50) | 30.6 (9.72) | 31.7 (8.86) | 32.4 (11.51) | 21.9 (3.44) | 30.2 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 7 | 6 | 4 | 31
  Male | 7 | 9 | 9 | 9 | 4 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 10 | 6 | 8 | 8 | 3 | 35
  Mixed Ethnic | 5 | 9 | 8 | 7 | 5 | 34
Weight [Mean (Standard Deviation); unit: kg] | 55.3 (8.58) | 55.9 (10.51) | 52.5 (9.82) | 53.5 (8.48) | 48.0 (8.70) | 53.6 (9.36)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 20.19 (4.031) | 20.09 (3.899) | 19.09 (2.562) | 19.41 (3.058) | 17.53 (1.785) | 19.43 (3.294)

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) Measured as the Daily Rate of Change in log10 CFUs (Colony Forming Units) of M. Tuberculosis in Sputum on Solid Media (Days 0-14).
Time Frame: Day 0 and Day 14
Population: Some of the EBA values could not be calculated due to missing results. The number of participants given are the number of participants for whom the results were available for this time period and therefore for whom the relevant EBA could be calculated.
Measure: Mean (Standard Deviation); unit: log10 CFU/ml
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 12 | 14 | 15 | 11 | 7
log10 CFU/ml | 0.106 (0.049) | 0.107 (0.053) | 0.091 (0.083) | 0.088 (0.084) | 0.148 (0.055)

2. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Daily Rate of Change in log10 CFUs (Colony Forming Units) of M. Tuberculosis in Sputum on Solid Media (Days 0-2).
Time Frame: Day 0 and Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU/ml
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 15 | 13 | 15 | 15 | 8
log10 CFU/ml | 0.109 (0.487) | 0.096 (0.226) | 0.025 (0.340) | -0.035 (0.420) | 0.403 (0.290)

3. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Daily Rate of Change in log10 CFUs (Colony Forming Units) of M. Tuberculosis in Sputum on Solid Media (Days 2-14).
Time Frame: Day 2 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU/ml
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 12 | 13 | 14 | 11 | 7
log10 CFU/ml | 0.106 (0.063) | 0.113 (0.079) | 0.095 (0.062) | 0.113 (0.099) | 0.112 (0.050)

4. Secondary Outcome: EBA Expressed as the Change in Time to Positive (TTP) Signal in Liquid Culture for M. Tuberculosis (Days 0-14)
Time Frame: Day 0 and Day 14
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 12 | 14 | 13 | 12 | 8
hours/day | 3.818 (2.327) | 4.776 (2.879) | 4.865 (3.461) | 4.440 (2.169) | 9.741 (5.249)

5. Secondary Outcome: EBA Expressed as the Change in Time to Positive (TTP) Signal in Liquid Culture for M. Tuberculosis (Days 0-2)
Time Frame: Day 0 and Day 2
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 13 | 13 | 11 | 15 | 8
hours/day | 1.115 (15.256) | 5.788 (12.173) | 2.795 (9.230) | 1.400 (7.659) | 24.125 (12.794)

6. Secondary Outcome: EBA Expressed as the Change in Time to Positive (TTP) Signal in Liquid Culture for M. Tuberculosis (Days 2-14) Show Description: [Not Specified]
Time Frame: Day 2 and Day 14
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Number analyzed (Participants) | 11 | 13 | 12 | 12 | 8
hours/day | 3.833 (2.954) | 5.09 (2.768) | 4.069 (1.916) | 4.868 (3.224) | 7.344 (4.66)

ADVERSE EVENTS:
Arm/Group | PA-824 200 mg | PA-824 600 mg | PA-824 1000 mg | PA-824 1200 mg | Rifafour
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/16 | 0/15 | 1/8
Other Adverse Events (participants affected / at risk) | 6/15 | 4/15 | 5/16 | 7/15 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PA-824 200 mg (N=15) | PA-824 600 mg (N=15) | PA-824 1000 mg (N=16) | PA-824 1200 mg (N=15) | Rifafour (N=8)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA-824 200 mg (N=15) | PA-824 600 mg (N=15) | PA-824 1000 mg (N=16) | PA-824 1200 mg (N=15) | Rifafour (N=8)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT corrected Interval Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in the Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — and Administration Site Conditions
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting, for review and removal of confidential information.